CLINICAL TRIAL: NCT06190184
Title: Testing the Efficacy of Viome Precision Supplements to Improve Clinical Outcomes for Mental Health Conditions
Brief Title: Viome Precision Nutritional Programs to Improve Clinical Outcomes for Mental Health Conditions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Viome (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V211.3.1
Record Dates: First submitted 2023-12-08; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Mental Health Issue; Mental Health Disorder; Mental Health; Depression; Depression, Anxiety; Anxiety; Anxiety Disorders; Anxiety Depression; Anxiety State
Keywords: Mental Health; diet; supplements; vitamins; stress
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, blinded, cohort study divided into two study arms: 1) control group (placebo), 2) precision-supplement
Who Masked: Participant
Masking Description: Once enrolled, participants are randomized into one of the 2 study arms. The coded supplements with blinded labels are shipped to the participants. The participants are not aware of which group they are randomized into.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants who have mental health issues are randomized into this study arm. They may be provided with any combination of nutritional recommendations and supplements. Placebo capsules will contain inert and inactive materials. Participants may need to use a mobile app in order to participate in the trial.
  Interventions: Other: Control arm
- Viome's Precision Nutrition Program (VPNP) (Experimental): Participants who have mental health issues are randomized into this study arm. They may be provided with any combination of nutritional recommendations and supplements. Participants may need to use a mobile app in order to participate in the trial.
  Interventions: Combination Product: VIOME Precision Nutrition Program

INTERVENTIONS:
Combination Product: VIOME Precision Nutrition Program — Precision supplement based on the participants microbiome sample results. Participants in this arm may have any combination of supplements, diet recommendations, and/or coaching.
  Other Names: VPNP
  Arms: Viome's Precision Nutrition Program (VPNP)
Other: Control arm — Participants who have mental health issues are randomized into this arm. They may be provided with any combination of nutritional recommendations and/or supplements. Placebo capsules will contain inert and inactive materials. Participants may need to use a mobile app in order to participate in the trial.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
US residents who have obesity and sign the informed consent form and are screened and enrolled for this study. Participants who are enrolled complete a survey upon enrollment and are randomized into one of two arms. This study is direct to participant and will not utilize clinical sites.

DETAILED DESCRIPTION:
Participants who meet the eligibility criteria are randomized into any of the two arms including: the placebo arm or the VIOME Precision Nutrition Program (VPNP) arm.

Placebo and Viome's Precision Nutrition Program include supplements and/or dietary recommendations towards improving the symptoms associated with metabolic wellness. The trial will last approximately 4 months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the United States
* 50 years old and older OR BMI of 25 or greater
* Able to speak and read English
* No unexplained weight loss, fevers, anemia, or blood in stool
* Willing and able to follow the trial instructions, as described in the recruitment letter
* Signed and dated informed consent prior to any trial-specific procedures.
* PHQ9 score of 5-24 (inclusive)

Exclusion Criteria:

* Unwilling to change their current diet
* Prior use of Viome products or services
* Antibiotic use in the previous 4 weeks
* Pregnancy (current or planned in the next 4 months)
* < 90 days postpartum
* Breast feeding
* Active infection
* Unable or unwilling to use Viome's App on an iPhone or Android smartphone
* Significant diet or lifestyle change in the previous 1 month
* IBD diagnosis -Major psychiatric/DSM-4 disease diagnosis (e.g. Schizophrenia, Bipolar disorder, Post- traumatic Stress Disorder, Obsessive Compulsive disorder)
* Use of investigational drugs, products or devices within 1 month prior to and 4 months after the start of the trial
* Cancer therapy within the previous 1 year
* Major surgery in the last 6 months or planned in the next 4 months
* Allergies to any supplement ingredients listed in the screening survey
* Currently on a specific diet: FODMAP, KETO, PALEO
* Answered yes to the question, "In the past few weeks, have you wished you were dead or had thoughts about killing yourself?"
* Gastrointestinal disease including:

  * GI surgery except:

    * Appendectomy and benign polypectomy
* Esophagitis
* Celiac disease
* GI malignancy or obstruction
* Peptic Ulcer Disease
* Duodenal or gastric ulcer disease

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in PHQ-9 Score | 4 months
  Change in PHQ-9 score for VPNP group compared to baseline scores.
Change in GAD-7 Score | 4 months
  Change in GAD-7 score for VPNP group compared to baseline scores.
Change in Quality of Life Score | 4 months
  Change in quality of life score for VPNP group compared to baseline scores.
Change in Perceived Stress Scale Score | 4 months
  Change in perceived stress score for VPNP group compared to baseline scores.

CONTACTS AND LOCATIONS:
Overall Officials: Momchilo Vuyisich, Principal Investigator — Viome
Locations (1):
- Viome Life Sciences, Bothell, Washington, United States